CLINICAL TRIAL: NCT02957578
Title: Post-Market Approval Study of the Solo Tympanostomy Tube Device
Brief Title: Clinical Study of Solo Tympanostomy Tube Device (TTD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: AventaMed DAC (Industry); University Hospitals of Derby and Burton NHS Foundation Trust (Other); Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13IH026; 208475 (Other: IRAS)
Record Dates: First submitted 2016-11-04; First posted 2016-11-07 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Otitis Media; Middle Ear Effusion
Keywords: Tympanostomy Tube; Ventilation Tube; Grommet; Otitis Media; Middle Ear Effusion
MeSH Terms: conditions — Otitis Media; Otitis Media with Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Solo TTD (Experimental): Placement of tympanostomy tube with Solo TTD
  Interventions: Device: Solo TTD

INTERVENTIONS:
Device: Solo TTD — Placement of tympanostomy tube with Solo TTD

SUMMARY:
This is a multi-centre, single arm study to evaluate the placement of tympanostomy tubes with the AventaMed Solo Tympanostomy Tube Device (TTD)

ELIGIBILITY:
Basic Inclusion Criteria:

* Listed for bilateral tympanostomy tube insertion only

Basic Exclusion Criteria:

* Anatomy that precludes sufficient visualisation of both the left and right eardrum with the Solo TTD in place.
* Anatomy that precludes safe access to both the left and right eardrum with the Solo TTD
* Patients in whom a reliable audiogram is not possible

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-09 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Device Success | Intraoperative
  Number of ears in which tube placement is achieved with the Solo TTD

SECONDARY OUTCOMES:
Conversion from moderate sedation | Intraoperative
  Number of patients requiring conversion from moderate sedation to general anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Owen Judd, Principal Investigator — Royal Derby Hospitals NHS Foundation Trust; Tawakir Kamani, Principal Investigator — Sheffield Children's NHS Foundation Trust; Matija Daniel, Study Chair — Nottingham University Hospitals NHS Trust; Anand Kasbekar, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No Plan to Share Individual Participant Data